CLINICAL TRIAL: NCT06609512
Title: A Clinical Study to Evaluate the Effect of Fasting Duration on the Pharmacokinetics of the Enlicitide in Healthy Adult Participants
Brief Title: A Clinical Study of Enlicitide and the Effect of Food in Healthy Adult Participants (MK-0616-033)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-033; MK-0616-033 (Other: MSD)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Enlicitide Treatment A (Experimental): Participants receive single oral dose of enlicitide after 8-hour overnight fast.
  Interventions: Drug: Enlicitide
- Enlicitide Treatment B (Experimental): Participants receive single oral dose of enlicitide 4 hours after morning meal.
  Interventions: Drug: Enlicitide
- Enlicitide Treatment C (Experimental): Participants receive single oral dose of enlicitide 3 hours after morning meal.
  Interventions: Drug: Enlicitide
- Enlicitide Treatment D (Experimental): Participants receive single oral dose of enlicitide 2 hours after morning meal.
  Interventions: Drug: Enlicitide

INTERVENTIONS:
Drug: Enlicitide — Oral Tablet
  Other Names: MK-0616; enlicitide decanoate

SUMMARY:
The goal of the study is to learn what happens to enlicitide decanoate in a healthy person's body over time when taken on an empty stomach or with food. Researchers will compare what happens to enlicitide in a healthy person's body over time when enlicitide is taken with or without food. Enlicitide decanoate will be referred to as "enlicitide" throughout.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has body mass index (BMI) ≥18 kg/m^2 and ≤32 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of gastrointestinal disease which may affect food and drug absorption, or has had a gastric bypass or similar surgery
* History of cancer (malignancy)
* Positive test(s) for Hepatitis B surface antigen (HBsAg), hepatitis C antibodies or Human immunodeficiency virus (HIV)
* History of a major surgery
* Is lactose intolerant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration versus Time Curve from 0 to Infinity (AUC0-inf) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  AUC0-inf of enlicitide in plasma will be determined.
Area Under the Concentration versus Time Curve from Time 0 to 24 hours (AUC0-24) of enlicitide in plasma | Pre-dose and at designated time points up to 24 hours post dose
  AUC0-24 of enlicitide in plasma will be determined.
Area under the concentration versus time curve from time 0 to last quantifiable sample (AUC0-last) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  AUC0-last of enlicitide in plasma will be determined.
Maximum plasma concentration (Cmax) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Cmax of enlicitide in plasma will be determined.
Time to maximum plasma concentration (Tmax) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Tmax of enlicitide in plasma will be determined.
Apparent terminal half-life (t1/2) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  t1/2 of enlicitide in plasma will be determined.
Apparent Clearance (CL/F) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  CL/F of enlicitide in plasma will be determined.
Apparent volume of distribution during terminal phase (Vz/F) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  Vz/F of enlicitide in plasma will be determined.
Lag Time (tlag) of enlicitide in plasma | Pre-dose and at designated time points up to 168 hours post dose
  tlag is the time from dosing to the first appearance in plasma. The tlag of enlicitide in plasma will be determined.

SECONDARY OUTCOMES:
Number of participants who experience one or more adverse events (AEs) | Up to ~ 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study intervention due to an AE | Up to ~ 14 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com